CLINICAL TRIAL: NCT06457685
Title: Pulse Intravascular Lithotripsy™ (Pulse IVL™) to Open Vessels With Calcific Walls and Enhance Vascular Compliance and Remodeling for Peripheral Artery Disease
Brief Title: Amplitude Vascular Systems (AVS) Lithotripsy POWER PAD 2 Trial
Acronym: POWER PAD 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amplitude Vascular Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-00005
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: PAD; Intravascular Lithotripsy; Lithotripsy; IVL; PAD II; PAD 2; Pulse IVL; Pulsatile Lithotripsy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, multicenter, non-randomized clinical study designed to demonstrate the safety and effectiveness of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy™ (Pulse IVL™) System for treatment of calcified (moderate to severe), stenotic, superficial femoral and popliteal arteries in patients with peripheral arterial disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pulse Intravascular Lithotripsy™ (Pulse IVL™) (Experimental): Pulse Intravascular Lithotripsy™ (Pulse IVL™) to open vessels with calcific walls
  Interventions: Device: Pulse Intravascular Lithotripsy (Pulse IVL)

INTERVENTIONS:
Device: Pulse Intravascular Lithotripsy (Pulse IVL) — The Pulse Intravascular Lithotripsy (Pulse IVL) System is used for the treatment of calcified (moderate to severe), stenotic, superficial femoral and popliteal arteries in patients with peripheral arterial disease.

SUMMARY:
POWER PAD 2 is a prospective, single-arm, multicenter, non-randomized clinical study designed to demonstrate the safety and effectiveness of the Amplitude Vascular Systems (AVS) Pulse Intravascular Lithotripsy™ (Pulse IVL™) System for treatment of calcified (moderate to severe), stenotic, superficial femoral and popliteal arteries in patients with peripheral arterial disease.

DETAILED DESCRIPTION:
POWER PAD 2 is a prospective, single-arm, multicenter, non-randomized clinical study designed to demonstrate the safety and effectiveness of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy™ (Pulse IVL™) System for treatment of calcified (moderate to severe), stenotic, superficial femoral and popliteal arteries in patients with peripheral arterial disease. This study will enroll subjects >18 years old that are presenting for a peripheral arterial disease intervention for the treatment of peripheral artery disease. Specifically, the subject has moderate to heavily calcified superficial femoral and popliteal arteries, presenting with Rutherford Category 2 to 4 of the target limb, with a reference vessel diameter (RVD) of 4mm to 6.5mm and a total lesion length of ≤ 150mm. Up to 120 subjects will be treated in the study at up to 20 U.S. investigational sites. Subjects will be evaluated at discharge, 30 days and 6 months after procedure.

ELIGIBILITY:
General Inclusion Criteria

Candidates will be included in the study only if all of the following conditions are met:

1. Able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
3. >18 years old
4. Rutherford Clinical Category 2, 3, or 4 of the target limb
5. Resting ankle-brachial index (ABI) of ≤0.90, or ≤0.75 after exercise, of the target leg OR ≥70% stenosis by prior imaging (CT/MR angiogram, DUS).
6. Subjects has de novo lesions who are felt to have indication for peripheral angiography and endovascular intervention by the investigator per their standard of care.
7. Estimated life expectancy >1 year, in the opinion of the investigator at the time of screening.

Angiographic Inclusion Criteria

Candidates will be included in the study only if all of the following intraoperative conditions are met:

1. Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guideline.
2. Target lesion that is located in a native de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to 2 cm above the bifurcation, or trifurcation, of the tibial artery).
3. Target lesion reference vessel diameter is between 4.0 mm and 6.5 mm by visual estimate.
4. Target zone is ≤ 150 mm in total contiguous treatable length. Target lesion can be all or part of the 150 mm zone.
5. Target lesion is ≥70% stenosis via visual estimate.
6. Subject has at least one patent tibial vessel on the target leg with runoff to the ankle (not supported by collateral circulation.) Tibial vessel patency is defined as no stenosis >50%.
7. Ability to pass the guidewire across the atherosclerotic lesion, without the use of re-entry devices.
8. No evidence of aneurysm or acute or chronic thrombus in target vessel.
9. Calcification is at least moderate. (Presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending ≥ 50% the length of the lesion.)

General Exclusion Criteria

Candidates will be excluded from the study if any of the following conditions are present:

1. Rutherford Clinical Category 0, 1, 5 and 6.
2. Active infection in the target leg.
3. Planned major amputation of the target leg (transmetatarsal or higher).
4. History of prior endovascular or surgical procedure on the target limb within the past 30 days.
5. Retrograde pedal/tibial access for intervention.
6. Known coagulopathy or has a bleeding diathesis, thrombocytopenia with platelet count < 100,000/microliter, or International Normalized Ratio (INR) >1.5.
7. Lesion in contralateral limb requiring intervention within the next 30 days.
8. Subject contraindicated for antiplatelet, anticoagulant, or thrombolytic therapy.
9. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
10. Known allergy to any Pulse IVL product materials.
11. Clinically significant myocardial infarction within 60 days prior to enrollment.
12. History of stroke within 60 days prior to enrollment.
13. History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to enrollment.
14. History of thrombolytic therapy within two weeks of enrollment.
15. Acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L), or on dialysis.
16. Pregnant or nursing.
17. Participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
18. Other medical, social, or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

Angiographic Exclusion Criteria

Candidates will be excluded from the study if any of the following intraoperative conditions are met:

1. The use of chronic total occlusion (CTO) re-entry devices.
2. Chronic Total Occlusion (CTO) greater than 40mm in length.
3. Any in-stent restenosis within the target zone.
4. Lesions within 10 mm of ostium of the SFA.
5. Highly tortuous arteries (bends greater than 30 degrees over the arc length of the balloon).
6. Target lesion within surgical bypass grafts.
7. Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract before target treatment zone (e.g. iliac or common femoral) not successfully treated without complications.
8. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to the target lesion at the time of the enrollment/index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Composite of New Onset Major Adverse Events (MAE) | Within 30-days of procedure
  MAE defined as experiencing any of the following: • The need for emergency surgical revascularization of target limb
  * Unplanned target limb amputation (above the ankle)
  * Symptomatic thrombus or distal emboli, defined as clinical signs or symptoms of thrombus or distal emboli detected in the treated limb in the area of the treated lesion, or distal to the treated lesion, after the index procedure and results in extended hospitalization or noted angiographically, and requiring mechanical or pharmacologic means to improve flow and results in extended hospitalization.
  * Perforations or dissections of grade D or greater that require an intervention such as bailout stenting.
Procedural Success | Time Frame: Day of procedure
  Defined as: The ability of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy (Pulse IVL) System to achieve a post Pulse IVL residual diameter stenosis of <50% (after adjunctive therapy, if used) as assessed by quantitative angiography via core lab evaluation.

SECONDARY OUTCOMES:
Device Success | Day of procedure
  The ability of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy (Pulse IVL) System to achieve a post Pulse IVL residual diameter stenosis of <50% (prior to adjunctive therapy) as assessed by quantitative angiography via core lab evaluation.
Clinical Success | Day of procedure
  The ability of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy (Pulse IVL) System to achieve a post Pulse IVL residual diameter stenosis of <50% (after adjunctive therapy, if used) as assessed by quantitative angiography via core lab evaluation and freedom from major adverse events that occur during the procedure.
Clinically Driven Target Lesion Revascularization | Within 30 days and six months of procedure
  Freedom from clinically driven target vessel revascularization as assessed by clinical presentation and diagnostic imaging.
Patency | Within 30 days and six months of procedure
  Target vessel patency by Duplex ultrasound, defined as freedom from > 50% restenosis, as assessed by Duplex ultrasound peak systolic velocity ratio of ≥2.5.
Technical Success | Day of procedure
  The ability of the Amplitude Vascular System (AVS) Pulse Intravascular Lithotripsy (Pulse IVL) System to deliver the Pulse IVL treatment to the desired location in the target vessel.
Ankle Brachial Index (ABI) | Within 30 days and six months of procedure
  Change in Ankle Brachial Index (ABI) of the target limb from baseline to follow-up
Walking Impairment Questionnaire (WIQ) | Within 30 days and six months of procedure
  Change in WIQ from baseline to follow-up
Freedom from major adverse events | Six months
  Freedom from major adverse events

OTHER OUTCOMES:
Prevalence of post-Pulse IVL Adjudicative Therapy | Day of procedure
  Prevalence of post-Pulse IVL Adjudicative Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Metzger, MD, Principal Investigator — Ohio Health
Locations (20):
- United States (20):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Vascular and Interventional Specialists of Orange County, Orange, California
  - Advanced Heart and Vein Center, Thornton, Colorado
  - Piedmont Heart Institute, Atlanta, Georgia
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Mercy Hospital South, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - Advanced Endovascular Physicians, West Orange, New Jersey
  - NYU Langone, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University and New York Presbyterian Hospital (NYPH), New York, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospital- Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside, Columbus, Ohio
  - Mainline Health Lankenau, Bryn Mawr, Pennsylvania
  - UPMC Pinnacle, Mechanicsburg, Pennsylvania
  - The Miriam Hospital - Brown University Health Partner, Providence, Rhode Island
  - Ascension Seton, Austin, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas